CLINICAL TRIAL: NCT01039428
Title: A Study of HS219 in Chronic Kidney Disease Patients on Hemodialysis With Hyperphosphatemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: KDL Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HS219CCR-001
Record Dates: First submitted 2009-12-24; First posted 2009-12-25 (Estimated); Results first posted 2012-06-01 (Estimated); Last update posted 2015-09-14 (Estimated); Status verified 2012-05

CONDITIONS: Hyperphosphatemia; Chronic Kidney Disease
Keywords: hyperphosphatemia; hemodialysis; chitosan
MeSH Terms: conditions — Hyperphosphatemia; Renal Insufficiency, Chronic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- HS219 (Experimental)
  Interventions: Dietary Supplement: HS219
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: HS219 — Chewing for 30 min three time a day far after meal
  Arms: HS219
Dietary Supplement: Placebo — Chewing for 30 min three times a day far after meal
  Arms: Placebo

SUMMARY:
This was a study to evaluate the efficacy and safety of HS219, chitosan-loaded chewing gum, when given three times a day for 3 weeks to the hemodialysis (HD) patients with hyperphosphatemia whose serum inorganic phosphorus was not well controlled with calcium carbonate or sevelamer hydrogen chloride.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent given
* Able to comply with the study procedures and medication
* On a stable HD regimen (at least 3 x per week) for ≥ 3 months
* Subject receiving calcium carbonate or sevelamer hydrochloride as a phosphate binder at screening, must have been on a stable regimen (dose and medication) for at least 1 month
* A mean serum inorganic phosphorous in the previous 3 tests : > 5.5 mg/dL and < 9.0 mg/dL
* Removal rate of blood urea nitrogen (BUN) ≥ 60%
* Rate of salivary flow by Saxon test ≥ 1 g/2 min

Exclusion Criteria:

* Blood purification therapy other than HD
* Current clinically significant intestinal motility disorder
* Possible parathyroid intervention during the study period
* History of malignancy and severe cardiovascular disorders such as heart disease, angina, congested heart failure, valve stenosis, atrial fibrillation and arrhythmia
* History of allergy against active ingredient
* Receipt of any investigational drug within 30 days of informed consent

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2009-12; Primary Completion 2010-05 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tadao Akizawa, MD, Study Chair — Divison of Nephrology, Department of Medicine, Showa University School of Medicine; Masafumi Fukagawa, MD, PhD, Study Director — Divison of Nephrology and Metabolism, Tokai University School of Medicine
Locations (11):
- Japan (11):
  - Meiyo Clinic, Toyohashi, Aichi-ken
  - Asahi General Hospital, Asahi, Chiba
  - Japanese Red Cross Koga Hospital, Koga, Ibaragi
  - Sumiyoshi Clinic Hospital, Mito, Ibaragi
  - Toride Medical Center, Toride, Ibaragi
  - Tsuchiura Kyodo General Hospital, Tsuchiura, Ibaragi
  - Japanese Red Cross Suwa Hospital, Suda, Nagano
  - Maruko General Hospital, Ueda, Nagano
  - Komagome Kyouritsu Clinic, Tokyo, Tokyo
  - Asagaya Suzuki Clinic, Tokyo, Tokyo
  - Suda Clinic, Tokyo, Tokyo

REFERENCES:
- [Derived] Natale P, Green SC, Ruospo M, Craig JC, Vecchio M, Elder GJ, Strippoli GF. Phosphate binders for preventing and treating chronic kidney disease-mineral and bone disorder (CKD-MBD). Cochrane Database Syst Rev. 2025 Jun 27;6(6):CD006023. doi: 10.1002/14651858.CD006023.pub4. PMID 40576086
- [Derived] Akizawa T, Tsuruta Y, Okada Y, Miyauchi Y, Suda A, Kasahara H, Sasaki N, Maeda Y, Suzuki T, Matsui N, Niwayama J, Suzuki T, Hara H, Asano Y, Komemushi S, Fukagawa M. Effect of chitosan chewing gum on reducing serum phosphorus in hemodialysis patients: a multi-center, randomized, double-blind, placebo-controlled trial. BMC Nephrol. 2014 Jun 25;15:98. doi: 10.1186/1471-2369-15-98. PMID 24968790

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Sixty eight HD patients maintained on calcium carbonate (33 subjects) or sevelamer (35 subjects) were enrolled during January - April, 2010. Sixty-three patients chewed at least one gum: 35 HS219 and 28 placebo.
Groups:
- HS219: Participants chewed HS219 chewing gum three times a day while fasting (i.e., between meals) for 30 min for 3 weeks.
- Placebo: Participants chewed placebo chewing gum three times a day while fasting (i.e., between meals) for 30 min for 3 weeks.
Period: Overall Study
Arm/Group | HS219 | Placebo
Started | 35 | 28
Completed | 33 | 28
Not Completed | 2 | 0
Not completed — Protocol Violation | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | HS219 | Placebo | Total
Number analyzed (Participants) | 35 | 28 | 63
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.1 (11.0) | 55.7 (11.3) | 56.4 (11.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 19 | 43
  Male | 11 | 9 | 20

OUTCOME MEASURES:

1. Primary Outcome: Change in Serum Inorganic Phosphorus at the End of Treatment From Baseline
Description: Change in serum inorganic phosphorus at the end of treatment from baseline
Time Frame: baseline and end of the chewing treatment during three week treatment period
Population: Full Analysis Set included all randomized participants who received at least one dose of study product. The endpoint was analyzed only for those participants who had data for this outcome measure.
Measure: Mean (Standard Deviation); unit: mg/dL
Groups:
- HS219: Participants chewed HS219 chewing gum for 30 min three times a day while fasting (i.e., between meals) for 3 weeks.
- Placebo: Participants chewed placebo chewing gum for 30 min three times a day while fasting (i.e., between meals) for 3 weeks.
Arm/Group | HS219 | Placebo
Number analyzed (Participants) | 35 | 28
mg/dL | -0.26 (1.19) | -0.20 (1.21)

2. Secondary Outcome: Number of Participants With Serum Inorganic Phosphorus Reduction of 1.5 mg/dL
Time Frame: baseline and end of the treatment
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | HS219 | Placebo
Number analyzed (Participants) | 35 | 28
participants | 7 [0.08 to 0.37] | 2 [0.01 to 0.24]

3. Secondary Outcome: Achievement Number of Participants With Serum Inorganic Phosphorus; 3.5 ≦P<5.5 mg/dL at Week 3
Time Frame: week 3
Population: Per Protocol Set included randomized participants who completed the entire clinical trial and were counted towards the final results. The endpoint was analyzed only for those participants who had data for this outcome measure.
Measure: Number; unit: participants
Arm/Group | HS219 | Placebo
Number analyzed (Participants) | 31 | 23
participants | 8 [0.12 to 0.45] | 2 [0.01 to 0.28]

4. Secondary Outcome: Serum Inorganic Phosphorus Level
Description: Serum inorganic phosphorus levels were determined at week 3 before the first dialysis of the week (Monday or Tuesday).
Time Frame: week 3
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | HS219 | Placebo
Number analyzed (Participants) | 33 | 28
mg/dL | 6.38 (1.35) | 6.29 (1.29)

5. Secondary Outcome: Salivary Inorganic Phosphorus Level
Description: Salivary inorganic phosphorus levels were determined at week 3 before the first dialysis of the week (Monday or Tuesday).
Time Frame: week 3
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | HS219 | Placebo
Number analyzed (Participants) | 32 | 28
mg/dL | 22.32 (8.04) | 21.51 (8.95)

6. Secondary Outcome: Corrected Serum Calcium (Ca) Level Based on the Serum Albumin Level Corrected Serum Calcium (mg/dL) = Measured Total Ca (mg/dL) + (4 - Serum Albumin [g/dL])
Description: Serum Ca levels were determined at week 3 before the first dialysis of the week (Monday or Tuesday).
Time Frame: week 3
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | HS219 | Placebo
Number analyzed (Participants) | 33 | 28
mg/dL | 9.37 (0.66) | 9.13 (0.61)

7. Secondary Outcome: Ca×P
Description: Serum inorganic phosphorus and Ca levels were determined at week 3 before the first dialysis of the week (Monday or Tuesday).
Time Frame: week 3
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mg/mL*mg/mL
Arm/Group | HS219 | Placebo
Number analyzed (Participants) | 33 | 28
mg/mL*mg/mL | 59.90 (13.87) | 57.24 (11.34)

8. Secondary Outcome: Serum Intact Parathyroid Hormone (PTH) Level
Description: Serum intact and whole PTH levels were determined at week 3 before the first dialysis of the week (Monday or Tuesday).
Time Frame: week 3
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | HS219 | Placebo
Number analyzed (Participants) | 33 | 28
pg/mL | 206.5 (141.2) | 251.2 (183.6)

9. Secondary Outcome: Serum Intact Fibroblast Growth Factor (FGF) 23 Level
Description: Serum intact FGF23 levels were determined at week 3 before the first dialysis of the week (Monday or Tuesday).
Time Frame: week 3
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: log10(pg/mL)
Arm/Group | HS219 | Placebo
Number analyzed (Participants) | 33 | 28
log10(pg/mL) | 4.0 (0.5) | 4.0 (0.5)

ADVERSE EVENTS:
Arm/Group | HS219 | Placebo
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/28
Other Adverse Events (participants affected / at risk) | 6/35 | 12/28
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HS219 (N=35) | Placebo (N=28)
common cold (Infections and infestations) | 4 (21) | 2 (10)
queasy (Gastrointestinal disorders) | 2 (21) | 10 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less